CLINICAL TRIAL: NCT03083145
Title: Evaluating How Breakfast Protein Source Affects Satiety, Glucose and Food Preference
Brief Title: Protein Source, Nutrition Messaging, and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Principal Investigator, Jamie Baum, Assistant Professor, University of Arkansas, Fayetteville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 15-05-753
Record Dates: First submitted 2017-03-09; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Messaging (Active Comparator): Whey protein beverage and pea protein beverages administered in a randomized order with a one- to two-week washout period between beverages.
  Interventions: Dietary Supplement: Whey Protein Beverage; Dietary Supplement: Pea Protein Beverage; Behavioral: Snack Tray Choices
- No Messaging (Active Comparator): Whey protein beverage and pea protein beverages administered in a randomized order with a one- to two-week washout period between beverages.
  Interventions: Dietary Supplement: Whey Protein Beverage; Dietary Supplement: Pea Protein Beverage; Behavioral: Snack Tray Choices

INTERVENTIONS:
Dietary Supplement: Whey Protein Beverage — Beverage administered and postprandial appetite assessed for 2 hours followed by 1 hour monitoring of food intake from ad libitum snack tray.
Dietary Supplement: Pea Protein Beverage — Beverage administered and postprandial appetite assessed for 2 hours followed by 1 hour monitoring of food intake from ad libitum snack tray.
Behavioral: Snack Tray Choices — Items were selected from a snack tray filled with healthy and unhealthy snacks in order to determine if educational messaging influenced snack choices. Shack choices wre recorded on a check list by a third party observer.

SUMMARY:
The objective of this study is to determine how the protein source and the physical form of food consumed at breakfast impact food intake. Research will be conducted by assessing feelings of hunger, food preference and blood glucose in healthy adults following the ingestion protein-based (animal versus plant) drinks similar calorie and protein content.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, no known health conditions

Exclusion Criteria:

* Taking medication, excluding hormonal birth control
* Food allergies
* Food intolerances

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Appetite assessment | 2 hours
  Appetite was assessed using visual analog scales

SECONDARY OUTCOMES:
Snack intake using checklist | 1 hour
  Snacks were provided after 2 hours and type and quantity of snacks consumed were monitored and recorded on a checklist by a member of the research team. At the end of the snacking period, uneaten portions of snacks were weighed and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No